CLINICAL TRIAL: NCT04041856
Title: Povidone-iodine 2% Eye Drop Versus Artificial Tear Drop for Treatment of Adenoviral Keratoconjunctivitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Farabi Eye Hospital (Other)
Responsible Party: Principal Investigator, mohammad soleimani, Associate professor of ophthalmology, Farabi Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: farabieyehospital
Record Dates: First submitted 2019-07-24; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Adenoviral Keratoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EKC patients (Active Comparator): Povidone-iodine 2% eye drop will be prescribed four times a day All patients will learn how to improve the hygiene level in order to reduce transmission
  Interventions: Drug: Povidone Ophthalmic
- Control group (No Intervention): All patients will undergo observational treatments including artificial tear drop and improving hygiene level

INTERVENTIONS:
Drug: Povidone Ophthalmic — Povidone-iodine 2% eye drop versus artificial tear drop for treatment of adenoviral keratoconjunctivitis
  Other Names: Povidone-iodine 2%
  Arms: EKC patients

SUMMARY:
Povidone-iodine 2% eye drop versus artificial tear drop for treatment of adenoviral keratoconjunctivitis

DETAILED DESCRIPTION:
Diagnosed EKC patients will be devided into two groups,first group will undergo povidone-iodine 2% eye drop four times a day and the control group will be treated only by artificial tear drops,they will be examined 3 months later and evaluations and data collections for the final comparison will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected for viral conjunctivitis

Exclusion Criteria:

* Allergic to iodized materials
* Age under 17

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-23 (Estimated); Primary Completion 2019-10-22 (Estimated); Study Completion 2019-11-22 (Estimated)

PRIMARY OUTCOMES:
Povidone-iodine 2% eye drop versus artificial tear drop for treatment of adenoviral keratoconjunctivitis | 3 months
  Decreased patient's symptoms
Povidone-iodine 2% eye drop | 3 months
  Decreased viral load based on PCR results